CLINICAL TRIAL: NCT04495114
Title: Pre-operative Carbohydrate Loading Patients With Diabetes Undergoing Elective Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RES0034025
Record Dates: First submitted 2020-07-23; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Modern fasting guidelines without the carbohydrate load preoperatively.
- Intervention Arm (Experimental): 40g carbohydrate load preoperatively.
  Interventions: Other: 40g carbohydrate load (Apple juice)

INTERVENTIONS:
Other: 40g carbohydrate load (Apple juice) — A 40g carbohydrate drink will be administered to subjects with non-insulin dependent type 2 diabetes 3 hours prior to their operation. This is standard practice in subjects without diabetes.
  Arms: Intervention Arm

SUMMARY:
Goal to evaluate the feasibility of conducting a large study that would assess the safety of carbohydrate drinks (i.e. juice) prior to elective colorectal surgery in patients with type 2 diabetes.

Traditionally, prior to surgeries involving general anesthetic, patients have been told not to eat or drink anything after midnight due to the risk of aspiration. More recent research have shown that it is safe to have clear fluids up to 2 hours before an operation and this is reflected in the current anesthesia clinical guidelines.

It is currently not known if it is safe for patients with type 2 diabetes to have a sugar drink before their surgery since they have trouble processing sugars and a subset of patients with diabetes are at increased risk to aspiration due to delayed gastric emptying.

DETAILED DESCRIPTION:
Fasting prior to the administration of a general anesthetic has been the standard of peri-operative care for many years. The refrain of "nothing to eat or drink after midnight" has become synonymous with surgery for both clinicians and the general public. The rationale behind this practice has been to reduce the risk of regurgitation of gastric contents. In addition, this instruction is straightforward for patients and ancillary staff, and allows for easy alteration of the order of cases on the operative list. Despite the widespread nature of this practice, a 2003 Cochrane review attempted to define the optimum duration of fasting, type of fasting, and volume of intake permitted and concluded that there was no evidence to suggest a shortened fluid fast resulted in an increased risk of aspiration, regurgitation, or morbidity in healthy patients.

Pre-operative fasting leads to insulin resistance and metabolic stresses. More recently it has been suggested that a preoperative carbohydrate loading may alleviate some deleterious effects of this fast. This strategy, combined with a number of others, have been recently introduced in many Enhanced Recovery After Surgery (ERAS) programs, that have led to improved postoperative pain, faster restoration of GI function, decreased LOS and decreased complication rate after colon surgery.

Type 2 diabetes is a disease of impaired glucose tolerance. It is a common condition that affects over 15% of general surgical patients undergoing major abdominal surgery. It is well recognized that this is a high-risk surgical population that is at increased risk of perioperative complications such as anastomotic dehiscence, poor wound healing, and postoperative ileus which can lead to an increased LOS after surgery. However, there is a relative dearth of robust evidence regarding preoperative fasting in patients with type 2 diabetes so there is no consensus among professional association guidelines internationally on recommendations for carbohydrate loading in this population undergoing elective surgery. Two major concerns have been raised; first the risk of aspiration in diabetic patients with a significant neuropathy and gastroparesis, and second potential for hyperglycemia and its deleterious effects.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, non-insulin dependent.
* Elective colorectal surgery patient at the University of Alberta Hospital, Grey Nuns Hospital, Misericordia Hospital, Foothills Hospital, or Royal Alexandra Hospital.

Exclusion Criteria:

* Insulin dependent type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Preoperative glucose | 1 to 2 hours prior to operation time.
  Mean difference in preoperative glucose between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Haili Wang, MD, Principal Investigator — Alberta Health services
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR